CLINICAL TRIAL: NCT06229145
Title: A Phase 4, Randomized, Double-blind, Multicenter Non-inferiority Trial Evaluating the Efficacy and Safety of Intravenous KRYSTEXXA® (Pegloticase) Administered Every 4 Weeks Compared With KRYSTEXXA Administered Every 2 Weeks With Co-administration of Weekly Doses of Methotrexate, Followed by an Open-label Extension, in Participants With Uncontrolled Refractory Gout (FORWARD II)
Brief Title: A Trial to Investigate the Non-inferiority of Pegloticase Administered Every 4 Weeks (Q4W) With MTX Compared With Every 2 Weeks (Q2W) With MTX in Participants With Uncontrolled Refractory Gout
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HZNP-KRY-409
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Gout
Keywords: Uncontrolled Gout; pegloticase; Krystexxa; Methotrexate; Chronic Gout
MeSH Terms: conditions — Gout | interventions — Pegloticase; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pegloticase + Methotrexate Q4W (Experimental): 16 mg pegloticase will be administered intravenously every 4 weeks for 24 weeks during double blind treatment and 24 weeks during open label.
  Interventions: Biological: Pegloticase; Drug: Methotrexate
- Pegloticase + Methotrexate Q2W (Experimental): 8 mg pegloticase will be administered intravenously every 2 weeks for 24 weeks during double blind treatment and 16 mg pegloticase every 4 weeks for 24 weeks during open label.
  Interventions: Biological: Pegloticase; Drug: Methotrexate

INTERVENTIONS:
Biological: Pegloticase — IV infusion
  Other Names: Krystexxa
Drug: Methotrexate — Oral

SUMMARY:
The study consists of 24-week double-blind trial to evaluate the non-inferiority of the efficacy and safety of pegloticase Q4W with MTX versus pegloticase Q2W with MTX, followed by a 24-week open-label extension of pegloticase Q4W with MTX, in participants with uncontrolled refractory gout.

The main objective of the study is to evaluate the effect of pegloticase 16 mg administered Q4W with MTX versus pegloticase 8 mg administered Q2W with MTX, on the response rate during Month 6, as measured by the sustained normalization of sUA to < 6 mg/dL for at least 80% of the time.

DETAILED DESCRIPTION:
Acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Adult men or women ≥ 18 years of age
2. Uncontrolled gout, defined as meeting the following criteria:

   * Hyperuricemia during the Screening Period, defined as sUA ≥ 7 mg/dL, and;
   * Failure to maintain normalization of sUA with xanthine oxidase inhibitors at the maximum medically appropriate dose, or with a contraindication to xanthine oxidase inhibitor therapy based on medical record review or participant interview, and;
   * Symptoms of gout
3. Willing to discontinue any oral ULT for at least 7 days prior to MTX dosing at Week -4 and continue not receiving any oral ULT when receiving pegloticase/placebo for pegloticase infusions
4. Women of childbearing potential must have negative serum/urine pregnancy tests during screening and Week -4.
5. Men who are not vasectomized must agree to use appropriate contraception, so as to not impregnate a female partner of reproductive potential during the trial.

Exclusion Criteria:

1. Severe chronic or recurrent bacterial infections, such as recurrent pneumonia or chronic bronchiectasis
2. Current or chronic treatment with systemic immunosuppressive agents, such as MTX, azathioprine or mycophenolate mofetil; prednisone > 10 mg/day or equivalent dose of other corticosteroid on a chronic basis (3 months or longer)
3. History of any transplant surgery requiring maintenance immunosuppressive therapy
4. Known history of hepatitis B virus surface antigen positivity or hepatitis B DNA positivity
5. Known history of hepatitis C virus RNA positivity, unless treated and viral load is negative
6. Known history of human immunodeficiency virus (HIV) positivity
7. G6PD deficiency (quantitative test at the Screening Visit centrally or locally)
8. Non-compensated congestive heart failure or hospitalization for congestive heart failure within 3 months of the Screening Visit, uncontrolled arrhythmia, treatment for acute coronary syndrome (myocardial infarction or unstable angina) or uncontrolled blood pressure (> 160/100 mmHg) prior to Week -4
9. Pregnant, planning to become pregnant, breastfeeding, planning to impregnate female partner or not on an effective form of birth control, as determined by the Investigator
10. Prior treatment with pegloticase, another recombinant uricase (rasburicase) or concomitant therapy with a PEG-conjugated drug
11. Unable to tolerate MTX 15 mg orally during the MTX Run-in Period
12. Chronic liver disease
13. White blood cell count < 4,000/μL, hematocrit < 32% or platelet count < 75,000/μL
14. Currently receiving systemic or radiologic treatment for ongoing cancer
15. History of malignancy within 5 years other than non-melanoma skin cancer or in situ carcinoma of cervix
16. Diagnosis of osteomyelitis
17. Known history of hypoxanthine-guanine phosphoribosyl-transferase deficiency, such as Lesch-Nyhan and Kelley-Seegmiller syndrome
18. A known intolerance to all protocol-standard gout flare prophylaxis regimens (i.e., participant must be able to tolerate at least 1 of the following: colchicine and/or non-steroidal anti-inflammatory drugs and/or low-dose prednisone ≤ 10 mg/day)
19. Current pulmonary fibrosis, bronchiectasis or interstitial pneumonitis. If deemed necessary by the Investigator, a chest X-ray may be performed during Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of pegloticase 16 mg administered Q4W with MTX versus pegloticase 8 mg administered Q2W with MTX, on the response rate as measured by the sustained normalization of sUA to < 6 mg/dL for at least 80% of the time | Month 6
  Proportion of participants achieving and maintaining serum uric acid (sUA) < 6 mg/dL at least 80% of the time

SECONDARY OUTCOMES:
Evaluate the effect of pegloticase 16 mg Q4W with MTX compared with pegloticase 8 mg Q2W with MTX on tophi resolution | Week 24
  Proportion of Participants with complete resolution of ≥ 1 tophus in participants with tophi at Baseline

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (74):
- United States (74):
  - The University of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Orthopedic Physicians Alaska - Rheumatology and Infusion, Anchorage, Alaska
  - Arizona Arthritis and Rheumatology Associates - Chandler, Chandler, Arizona
  - Arizona Arthritis and Rheumatology Rese, Flagstaff, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Gilbert, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Mesa, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - Arizona Arthritis and Rheumatology Research, Phoenix, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Sun City, Arizona
  - Arizona Arthritis and Rheumatology, Tucson, Arizona
  - Covina Arthritis Clinic, Covina, California
  - Medvin Clinical Research- Riverside, Hemet, California
  - Velocity Clinical Research - Boise - ERN - PPDS, North Hollywood, California
  - TriWest Research Associates, San Diego, California
  - Precision Comprehensive Clinical Research Solutions, San Leandro, California
  - Saint John's Health Center - Providence St John's Health Ctr, Santa Monica, California
  - C.V. Mehta MD Medical Corporation, Temecula, California
  - Foothill Arthritis, Tujunga, California
  - Medvin Clinical Research, Whittier, California
  - University of Colorado Denver, Aurora, Colorado
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Denver Arthritis Clinic - Rheumatology, Denver, Colorado
  - Arthritis & Rheumatic Disease, Aventura, Florida
  - Prohealth Research Center, Doral, Florida
  - Life Clinical Trials, Margate, Florida
  - Homestead Associates in Research,Inc, Miami, Florida
  - D&H National Research Centers, Inc., Miami, Florida
  - Well Pharma, Miami, Florida
  - Felicidad Medical Research, LLC., Miami, Florida
  - New Generation Of Medical Research, Naples, Florida
  - IRIS Research & Development, Plantation, Florida
  - D&H Pompano Research Center, Pompano Beach, Florida
  - D&H Tamarac Research Center, Tamarac, Florida
  - GCP Clinical Research, Tampa, Florida
  - ClinPro Research Solutions, LLC, Tampa, Florida
  - Arthritis Center of North Georgia, Gainesville, Georgia
  - Vista Clinical Research, LLC, Newnan, Georgia
  - Great Lakes Clin. Trials, Chicago, Illinois
  - Conquest Research - Anesthesiology/Pain Medicine, Chicago, Illinois
  - Great Lakes Clinical Trials - Gurnee, Highland Park, Illinois
  - Crowley CORE - Illinois Bone and Joint Institute, Hinsdale, Illinois
  - Lake Cumberland Rheumatology, PLLC, New Albany, Indiana
  - L-MARC Research Center, Louisville, Kentucky
  - Velocity CR - New Orleans, Covington, Louisiana
  - Velocity CR - New Orleans, New Orleans, Louisiana
  - Michigan Medicine, Ann Arbor, Michigan
  - June DO,PC, Lansing, Michigan
  - Clinical Research Institute of Michigan, LLC, Saint Clair Shores, Michigan
  - Inspire Santa Fe Medical Group, Santa Fe, New Mexico
  - Velocity Clinical Research-Vestal, Vestal, New York
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - Research Carolina Elite, Denver, North Carolina
  - Triad Clinical Trials - Gastroenterology, Greensboro, North Carolina
  - Accellacare of Hickory, Hickory, North Carolina
  - Cape Fear Arthritis Care, Leland, North Carolina
  - Shelby Clinical Research - Family Medicine, Shelby, North Carolina
  - Velocity Clinical Research- Cincinatti, Cincinnati, Ohio
  - Velocity Clinical Research - Cleveland, Cleveland, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Velocity Clinical Research, Spartanburg - Pulmonology, Greenville, South Carolina
  - Premier Clinics Pa - Rock Hill, Sc, Rock Hill, South Carolina
  - Low Country Rheumatology, Summerville, South Carolina
  - Amarillo Center for Clinical Research, Ltd., Amarillo, Texas
  - Clinical Trial Network, Austin, Texas
  - Synergy Groups Medical LLC, Houston, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - AIM Trials - Internal Medicine, Plano, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Texas Research Center, Sugar Land, Texas
  - Velocity Clinical Research - Salt Lake City (West Jordan), West Jordan, Utah
  - Velocity Clinical Research-Portsmouth, Portsmouth, Virginia
  - Arthritis Northwest, PLLC - Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com